CLINICAL TRIAL: NCT04221737
Title: Early Use of Airway Pressure Release Ventilation (APRV) in Patients With Acute Respiratory Distress Syndrome
Brief Title: Early Use of Airway Pressure Release Ventilation (APRV) in ARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Miguel Á Ibarra-Estrada, Principal investigator, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCG/CEI-0632/17
Record Dates: First submitted 2020-01-05; First posted 2020-01-09 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; Acute Lung Injury; Mechanical Ventilation; APRV
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional ventilation (Active Comparator): Protective lung conventional strategy with volume-controlled ventilation (VCV) or pressure-controlled ventilation (PCV) mode, with low tidal volume and adequate positive end expiratory pressure (PEEP) level.
  Interventions: Device: Conventional. General Electric Healthcare Engstrom ventilator system
- Time-controlled adaptive APRV (Experimental): Airway Pressure Release Ventilation with Time-controlled adaptive ventilation method. Allowing for spontaneous breathing.
  Interventions: Device: APRV. General Electric Healthcare Engstrom ventilator system

INTERVENTIONS:
Device: APRV. General Electric Healthcare Engstrom ventilator system — APRV consist of an extended time at plateau pressure (a continuous positive airway pressure phase) comprising about 90% of the respiratory cycle, while providing very brief releases to enhance carbon dioxide removal. Time-controlled adaptive method requires interpretation of the expiratory flow curve to assess changes in lung elastance and, therefore, set the Time low to optimize carbon dioxide removal, but not at the expense of alveolar derecruitment and instability.
  Arms: Time-controlled adaptive APRV
Device: Conventional. General Electric Healthcare Engstrom ventilator system — Lung protective ventilation consist of delivery of low tidal volumes (4-6 ml/kg PBW), high PEEP enough to avoid de-recruitment, titrated according to ARDSNet PEEP/fraction of inspired oxygen (FiO2) table, while avoiding excessive transpulmonary pressure.
  Arms: Conventional ventilation

SUMMARY:
Airway pressure release ventilation (APRV) is a time-cycled, pressure controlled, intermittent mandatory ventilation mode with extreme inverse I:E ratios. Currently it is considered as a non-conventional ventilatory mode. The investigators aim to compare APRV with conventional mechanical ventilation (MV) in patients with acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
Despite the advances in technology and ventilatory modes, mortality of ARDS is still around 40%. Besides prone positioning, the best approach of management is low tidal volume ventilation (LTV). This 'protective ventilation' strategy is not aways effective to improve oxygenation and is associated with an increased requirement of sedation and neuromuscular blocking agents, which increase length of stay and morbidity. APRV is a ventilatory mode based on relatively high and sustained continuous positive pressure, combined with a short phase of release to allow carbon dioxide removal. It also allows unrestricted spontaneous breathing throughout respiration, independent of the ventilator cycle. Providing sustained inflation while limiting duration and frequency of release phase permits limiting volume loss, resulting in progressive and improved alveolar recruitment, an increased alveolar surface area available for gas exchange and improved ventilation-perfusion matching.

In this multi-center, prospective, randomized, controlled, open trial, the investigators aim to compare the effects and safety of the early application of time-controlled adaptive method of APRV and conventional ventilation with LTV strategy in patients with severe to moderate ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory distress syndrome, according to the Berlin definition of ARDS, with adjusted pO2/FiO2 for altitude <300, and less than 48 h of endotracheal mechanical ventilation

Exclusion Criteria:

* Pregnancy
* Less than 18 years-old
* Expected duration of mechanical ventilation less than 48 h
* Preexisting conditions with an expected 3-month mortality exceeding 50%
* Concurrent chemotherapy
* Confirmed intracranial hypertension
* Catastrophic cranial trauma or neuromuscular disorders that are known to prolong mechanical ventilation
* Pneumothorax at enrollment (resolved or not)
* Do-not-resuscitate order

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-07-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation free days | 28 days

SECONDARY OUTCOMES:
All causes mortality | 28 days
ICU length of stay | 28 days
Hospital length of stay | 60 days
Mean airway pressure, peak airway pressure, maximum P high | 7 days
  Measured in cmH20
Average expiratory time | 7 days
  Measured in seconds
Minute ventilation | 7 days
oxygen partial pressure (pO2) | 7 days
pCO2 (carbon dioxide partial pressure) | 7 days
Mean arterial pressure | 7 days
Maximum dosage of vasopressors requirement | 7 days
Richmond Sedation-Agitation Scale | 7 days
  Range from -5 (unarousable) to +4 (combative)
Average dose of propofol use | 7 days
Rate of neuromuscular blocking agents utilization | 7 days
Prone position rate | 7 days
Average of prone position sessions | 7 days
Rate of recruitment maneuvers | 7 days
Tracheostomy rate | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ibarra-Estrada, Dr, Principal Investigator — Hospital Civil Fray Antonio Alcalde
Locations (1):
- Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez Saubidet I, Maskin LP, Rodriguez PO, Bonelli I, Setten M, Valentini R. Mortality in patients with respiratory distress syndrome. Med Intensiva. 2016 Aug-Sep;40(6):356-63. doi: 10.1016/j.medin.2015.10.007. Epub 2015 Dec 31. English, Spanish. PMID 26746127
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Albert S, Kubiak BD, Vieau CJ, Roy SK, DiRocco J, Gatto LA, Young JL, Tripathi S, Trikha G, Lopez C, Nieman GF. Comparison of "open lung" modes with low tidal volumes in a porcine lung injury model. J Surg Res. 2011 Mar;166(1):e71-81. doi: 10.1016/j.jss.2010.10.022. Epub 2010 Nov 12. PMID 21195426
- [Background] Sydow M, Burchardi H, Ephraim E, Zielmann S, Crozier TA. Long-term effects of two different ventilatory modes on oxygenation in acute lung injury. Comparison of airway pressure release ventilation and volume-controlled inverse ratio ventilation. Am J Respir Crit Care Med. 1994 Jun;149(6):1550-6. doi: 10.1164/ajrccm.149.6.8004312.
- [Derived] Ibarra-Estrada MA, Garcia-Salas Y, Mireles-Cabodevila E, Lopez-Pulgarin JA, Chavez-Pena Q, Garcia-Salcido R, Mijangos-Mendez JC, Aguirre-Avalos G. Use of Airway Pressure Release Ventilation in Patients With Acute Respiratory Failure Due to COVID-19: Results of a Single-Center Randomized Controlled Trial. Crit Care Med. 2022 Apr 1;50(4):586-594. doi: 10.1097/CCM.0000000000005312. PMID 34593706